CLINICAL TRIAL: NCT04786613
Title: The Efficacy and Safety of Intra-articular Injections of 48 mg, 32 mg and 20 mg Linear Hyaluronic Acid in Patients With Knee Osteoarthritis: A Multicenter Randomized Single-Blind Clinical Trial
Brief Title: The Effectiveness of Different Doses of Hyaluronic Acid Injections in Knee Osteoarthritis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Selim Sezikli, MD, Sub-Investigator, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Istanbul University HA
Record Dates: First submitted 2021-03-03; First posted 2021-03-08 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Osteoarthritis; Linear Hyaluronic Acid
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 20 mg, 1.0% hyaluronic acid injection groups (Active Comparator): In the first group, 2 ml linearly linked 20 mg 1.0% hyaluronic acid injection in 5 sessions will be applied.
  Interventions: Other: Intra-articular 20 mg, 1.0% Hyaluronic Acid Injection
- 32 mg, 1.6% hyaluronic acid injection groups (Active Comparator): In the second group, 2 ml linearly linked 32 mg 1.6% hyaluronic acid injection in 3 sessions will be applied.
  Interventions: Other: Intra-articular 32 mg, 1.6% Hyaluronic Acid Injection
- 48 mg, 2.0% hyaluronic acid injection groups (Active Comparator): In the third group 2.4 ml linearly linked 48 mg 2.0% hyaluronic acid injection in a single sessions will be applied.
  Interventions: Other: Intra-articular 48 mg, 2.0% Hyaluronic Acid Injection

INTERVENTIONS:
Other: Intra-articular 20 mg, 1.0% Hyaluronic Acid Injection — Intra-articular 2 ml linearly linked 20 mg 1.0% hyaluronic acid injection in 5 sessions will be applied.
  As a home exercise program, hamstring and quadriceps stretching, quadriceps isometric strengthening, short arc terminal extension exercises will be given at least three days a week with 3 sets of 10 repetitions.
  Arms: 20 mg, 1.0% hyaluronic acid injection groups
Other: Intra-articular 32 mg, 1.6% Hyaluronic Acid Injection — Intra-articular 2 ml linearly linked 32 mg 1.6% hyaluronic acid injection in 3 sessions will be applied.
  As a home exercise program, hamstring and quadriceps stretching, quadriceps isometric strengthening, short arc terminal extension exercises will be given at least three days a week with 3 sets of 10 repetitions.
  Arms: 32 mg, 1.6% hyaluronic acid injection groups
Other: Intra-articular 48 mg, 2.0% Hyaluronic Acid Injection — Intra-articular 2,4 ml linearly linked 48 mg 2.0% hyaluronic acid injection in single session will be applied.
  As a home exercise program, hamstring and quadriceps stretching, quadriceps isometric strengthening, short arc terminal extension exercises will be given at least three days a week with 3 sets of 10 repetitions.
  Arms: 48 mg, 2.0% hyaluronic acid injection groups

SUMMARY:
The aim of this prospective, randomized, controlled multi-centre study is to compare the effectiveness and safety of three and five injections of standard linear hyaluronic acid (HA) versus single HA injection in terms of pain intensity and functional status in patients with knee osteoarthritis.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is the most common form of chronic joint disease. A treatment option for patients diagnosed with knee osteoarthritis is intra-articular hyaluronic acid therapy. In this prospective, randomized controlled, single blind, interventional study, a total of 90 patients with stage 2-3 knee osteoarthritis according to the kellgren lawrence classification who meet the eligibility criteria will be enrolled in the study. Eligible participants will be randomly assigned to one of the three groups using computer-generated random numbers. In the first group, 2 ml linearly linked 20 mg 1.0% hyaluronic acid injection in 5 sessions, in the second group 2 ml linearly linked 32 mg 1.6% hyaluronic acid injection in 3 sessions and in the third group 2.4 ml linearly linked 48 mg 2.0% hyaluronic acid injection in a single sessions will be applied. Participants are going to evaluate before injection, at the 1-month follow-up, at the 3-month follow-up and 6-month follow-up using the visual analog scale (VAS) scores for pain during activity, at rest, and at night, with the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) change in pain, stiffness and physical function score, the change in the Timed Up and Go Test (TUG) time and the change in the patient's daily activities with the numerical global patient assessment scale.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral or bilateral symptomatic knee pain for at least three months
* Presence of Kellgren-Lawrence stage 2-3 osteoarthritis on current anterior-posterior knee radiographs
* Functional ambulation scale stage 4-5
* Being able to attend injection and control examinations

Exclusion Criteria:

* Intra-articular knee injection within the last six months
* History of severe trauma to the knee within the past six months
* Concomitant severe meniscus or ligament injury, surgery applied to the knee area
* Presence of severe effusion, inflammatory joint disease, infection, hematological and oncological disease in the knee.
* Having a bleeding disorder and / or using warfarin
* Kellgren-Lawrence stage 1 or stage 4 osteoarthritis on current anterior-posterior knee radiographs
* Presence of cardiac or systemic disease that may affect exercise
* The presence of neurological disease and psychiatric disease such as Parkinson's disease, stroke history that may affect balance
* Body Mass Index ≥35 kg / m²
* Allergy to hyaluranic acid products

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2021-10-07 (Actual); Study Completion 2021-11-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline activity pain score at 1-months, 3-months and 6-months | Baseline, 1-month, 3-month, 6-month
  Visual Analogue Scale-Activity pain (0-10 point). Higher scores mean a worse outcome

SECONDARY OUTCOMES:
Change from baseline rest pain score at 1-months, 3-months and 6-months | Baseline, 1-month, 3-month, 6-month
  Visual Analogue Scale-Rest pain (0-10 point). Higher scores mean a worse outcome
Change from baseline night pain score at 1-months, 3-months and 6-months | Baseline, 1-month, 3-month, 6-month
  Visual Analogue Scale-Night pain (0-10 point). Higher scores mean a worse outcome
Change from baseline pain, stiffness and physical function at 1-months, 3-months and 6-months | Baseline, 1-month, 3-month, 6-month
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) measures knee pain, stiffness, and physical function. The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. The sum of the scores for the three subscales gives a total WOMAC score. High scores are associated with more pain, stiffness, and poor function, while low scores indicate well-being.
Change from baseline functional balance at 1-months, 3-months and 6-months | Baseline, 1-month, 3-month, 6-month
  The Timed Up and Go test requires the person to stand up from a standard chair in which they are sitting, walk 3 m at a comfortable speed to the marked place on the floor, turn around, walk backwards to the starting point and return to the sitting position in the chair. The time taken for the person to complete the test is measured in seconds. The timing of the test is related to the function.

CONTACTS AND LOCATIONS:
Overall Officials: Demirhan Diracoglu, Prof., Principal Investigator — Istanbul University Istanbul Faculty of Medicine, Department of Physical Medicine and Rehabilitation
Locations (1):
- Istanbul University Istanbul Faculty of Medicine, Department of Physical Medicine and Rehabilitation, Istanbul, Fatih, Turkey (Türkiye)